CLINICAL TRIAL: NCT01723371
Title: Beta Blockers for Treatment of Pulmonary Arterial Hypertension in Children
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of enrollment.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Friedberg, Staff Cardiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000031903
Record Dates: First submitted 2012-10-31; First posted 2012-11-07 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH; Pediatrics; Right Heart Failure (RHF); Carvedilol; Beta-blockers
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carvedilol (Experimental)
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will be administered orally. The initial dose of carvedilol will be 0.05mg/kg/day divided into 2 doses. After two weeks, at subsequent weekly study visits, the dose of carvedilol will be increased incrementally to 0.1mg/kg in Week 2, 0.2mg/kg in Week 3, 0.4mg/kg in Week 4, 0.6mg/kg in Week 5, and 0.8mg/kg in Week 6, when the target dose of 0.8mg/kg/day (if weight is less than 62.5kg) or 50mg/day (if weight is greater than 62.5kg) is achieved. This dosage, assuming no adverse effects, will be maintained between Weeks 6 and 30 of the study. After the maintenance period from Week 6 to 30, patients will be weaned over 5 to 7 days or continued on a non-study drug supply.

SUMMARY:
This study will determine the safety and feasibility of using a β-blocker (in this case carvedilol) in the treatment of pediatric patients with Left Heart Failure (LHF) in children with Pulmonary Arterial Hypertension (PAH). Carvedilol affects the nervous system, the same system that is highly activated in response to stress in patients with PAH. Each patient is administered a dosage of carvedilol, according to their weight. This dosage is increased incrementally over the span of the study, if the patient responds well to the drug. The study will determine whether the potential adverse side effects of carvedilol outweigh the possible positive results in reducing LHF. The hypothesis of this study predicts that carvedilol will have positive effects in treating LHF, similar to their use in treatment of Right Heart Failure (RHF). This is a single-centered pilot study. Each patient will be studied for approximately 31 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 8 and ≤ 17.5 years of age at the time of study enrollment.
* Patients must have a mean pulmonary artery pressure of greater than 25mmHg at rest in a setting of normal pulmonary arterial wedge pressure of 15mmHg or less with a PVR index greater than 3 Woods units•m2 at last hemodynamic study.
* Patients must be diagnosed with any of the following:Idiopathic PAH (IPAH), PAH associated with repaired congenital heart disease, PAH associated with minor congenital heart disease (small interventricular communication, small interarterial communication, small ductus arteriosis)
* Patients must be clinically stable (i.e. no treatment changes) for the last 3 months
* Patients must have no or minimal evidence of fluid overload or volume depletion judged by clinical evaluation (with or without diuretic treatment)
* Written informed consent

Exclusion Criteria:

* Patients who are unable to perform a six minute walk test (6MWT)
* Patients with a known history of pulmonary hypertension secondary to venoocclusive disease and/or capillary hemangiomatosis; pulmonary hypertensions owing to left heart disease
* Patients who have previously received treatment with an intravenous positive inotropic agent in the last 3 months
* Patients who are currently receiving β-blockers
* Patients with a known history of reactive airways disease (bronchial asthma or relate bronchospastic conditions)
* Patients with chronic obstructive pulmonary disease (COPD)
* Patients with a known history of adverse reaction to β-blockers
* Patients with a heart block on ECG or resting heart rate < 60 bpm
* Patients with systemic hypotension (below 5th percentile for age) are not eligible as follows: 1-10 years old: systolic blood pressure defined as < [70 + (2 x age in years)] mmHg; Older than 10 years: systolic blood pressure < 90 mmHg
* Patients with coagulopathy (INR < 1.5 or platelet count <50,000/mm3)
* Patients with a known history of severe hepatic impairment (defined by the presence of ascites, esophageal varices, jaundice or spider angiomata)
* Patients with severe renal insufficiency (defined as creatinine clearance < 30 mL/min/m2)
* Patients with a known malignancy or other co-morbidity expected to limit survival or to limit the ability to complete the study
* Patients with trisomy 21
* Patients with a known history of sick sinus syndrome
* Patients with a known history of moderate or severe primary obstructive valvular heart disease
* Patients with a known history of diabetes
* Female patients who are pregnant of breast-feeding

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Throughout study (Baseline to week 31)
  -Incidence of major adverse effects defined as bradycardia, hypotension, and syncope, worsening of symptoms, disease state and death

SECONDARY OUTCOMES:
Improvement in the six minute walk test (6MWT) and cardiopulmonary exercise testing (CPX) | Change over 6 months
  This will be measured by the difference in walking distance in the 6MWT and peak oxygen consumption in the CPX, between the baseline condition before the study and after 6 months with maintenance dose of carvedilol.
Improvement in echocardiogram and magnetic resonance imaging (MRI) parameters | Change over 6 months
  The echocardiogram will be a subjective assessment of the right valve (RV) fractional area of change through TAPSE. The MRI will measure the RV ejection fraction. Both indicators will measure the different between the baseline condition before the study and after 6 months with maintenance dose of carvedilol.
Feasibility of carvedilol | Baseline, Week 0, 2, 3, 4, 5, 6, 10, 18, 22, 30, 31
  * Proportion of patients achieving target maintenance dose of carvedilol
  * Proportion of patients requiring dose adjustment due to bradycardia and/or hypertension
  * Proportion of patients stopping treatment with carvedilol due to serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mark Friedberg, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada